CLINICAL TRIAL: NCT04445090
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 1569912 in Healthy Male Subjects (Single-blind, Partially Randomized Within Dose Groups, Placebo-controlled, Parallel-group Design) With an Additional Relative Bioavailability/ Food Effect Part (Open-label, Randomized, Three-way Crossover Design)
Brief Title: A Study in Healthy Men to Test How Well Different Doses of BI 1569912 Are Tolerated and How Food Influences the Amount of BI 1569912 in the Blood
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Identification of potential mutagenic metabolite in human plasma
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1447-0001; 2019-004836-51 (EudraCT Number)
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: SRD-Part: parallel-group design BA/FE-Part: three-way crossover design
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Rising Dose part: BI 1569912 (Experimental)
  Interventions: Drug: BI 1569912
- Single Rising Dose part: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Bioavailability and Food effect part: BI 1569912 (Experimental): This part follows the SRD part; open-label, randomised, single-dose, intraindividual, six-sequence, three-way crossover
  Interventions: Drug: BI 1569912

INTERVENTIONS:
Drug: BI 1569912 — BI 1569912
  Arms: Bioavailability and Food effect part: BI 1569912; Single Rising Dose part: BI 1569912
Drug: Placebo — Placebo
  Arms: Single Rising Dose part: Placebo

SUMMARY:
SRD-Part: To investigate safety, tolerability, pharmacokinetics and pharmacodynamics following single rising doses (SRD) of BI 1569912 BA/FE-Part: To investigate (a) the relative bioavailability (BA) of BI 1569912 and (b) the influence of food (FE) on the relative bioavailability of BI 1569912

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR), respiratory rate (RR), temperature (T)), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation
* Male subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods (of female partners) plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device
  * Sexually abstinent
  * Surgically sterilised (including hysterectomy of female partner)
  * Postmenopausal female partner, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular, hepatic parameters (alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin) or renal parameters (creatinine) exceeding the upper limit of normal (ULN) after repeated measurements
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* History of relevant orthostatic hypotension, fainting spells, or any unexplained blackouts
* Chronic or relevant acute infections
* A positive polymerase chain reaction (PCR) test for SARS-CoV-2/COVID-19 and/ or any clinical symptom suggestive for this disease at screening and on Day -3.

Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
SRD-part: % of subjects with drug-related adverse events | up to 14 days
BA/FE-part: AUC0-tz (area under the concentration-time curve of BI 1569912 in plasma over the time interval from 0 to the last quantifiable data point) | up to 4 days
BA/FE-part: Cmax (maximum measured concentration of BI 1569912 in plasma) | up to 4 days

SECONDARY OUTCOMES:
SRD-Part: AUC0-∞ (area under the concentration-time curve of BI 1569912 in plasma over the time interval from 0 extrapolated to infinity) | up to 4 days
SRD-Part: Cmax (maximum measured concentration of BI 1569912 in plasma) | up to 4 days
BA/FE-Part: AUC0-∞ (area under the concentration-time curve of BI 1569912 in plasma over the time interval from 0 extrapolated to infinity) | up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com